CLINICAL TRIAL: NCT04261504
Title: Brain Mechanisms of Reducing Polysubstance Use Following a Novel Body-mind Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB2018-943; R61AT010138 (NIH)
Record Dates: First submitted 2019-12-22; First posted 2020-02-07 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Multiple Drug Use

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrative Body Mind Training (IBMT) (Experimental): mindfulness
  Interventions: Behavioral: IBMT
- Relaxation Training (RT) (Active Comparator): relaxation
  Interventions: Behavioral: RT

INTERVENTIONS:
Behavioral: IBMT — mindful presence in a non-judgmental way
  Arms: Integrative Body Mind Training (IBMT)
Behavioral: RT — progressive muscle relaxation
  Arms: Relaxation Training (RT)

SUMMARY:
The proposed study will examine brain mechanisms of a brief mindfulness intervention - integrative body-mind training (IBMT) on alcohol, tobacco, and cannabis (ATC) reduction.

DETAILED DESCRIPTION:
The R61 phase of the proposed study will examine brain mechanisms of a brief mindfulness intervention - integrative body-mind training (IBMT) that targets at self-control networks in the brain, and test IBMT effects on alcohol, tobacco, and cannabis (ATC) reduction.

ELIGIBILITY:
Inclusion Criteria:

* (1) at least 18 years old;
* (2) free of any psychiatric diagnoses or medication (besides a substance use disorder to alcohol, tobacco, or cannabis);
* (3) in the past month, at least 4 episode of heavy episodic drinking; at least 3 occasion of cannabis use; and daily cigarette use for at least the past month;
* (4) normal or corrected-to-normal vision;
* (5) written informed consent;
* (6) no previous meditation or neurofeedback (NF) experiences.

Exclusion Criteria:

* (1) any psychiatric diagnoses other than a substance use disorder;
* (2) medical disorder(s) that may affect the central nervous system; medications that affect the central and autonomic nervous system; or a positive pregnancy test result (females);
* (3) excluding cannabis, evidence of recent (past month) illicit drug use.

Ages: 18 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-04-19 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Yuan Tang, Principal Investigator — Texas Tech University
Locations (1):
- TTU/UT, Lubbock, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integrative Body Mind Training (IBMT) | Relaxation Training (RT)
Started | 35 | 35
Completed | 30 | 28
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrative Body Mind Training (IBMT) | Relaxation Training (RT) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 18 | 17 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 24 | 24 | 48
  Hispanic or Latino | 11 | 11 | 22
  Unknown/Not Reported Ethnicity | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Brain Changes in Functional Activity
Description: 70 participants with polysubstance use are assessed by changes of brain in functional activity of anterior cingulate cortex before (baseline) and post-intervention (2 weeks).
Time Frame: The outcome measure is assessed at baseline and post-intervention.
Measure: Mean (Standard Deviation); unit: beta weights
Arm/Group | Integrative Body Mind Training (IBMT) | Relaxation Training (RT)
Number analyzed (Participants) | 30 | 28
beta weights
  Baseline | 0.7 (1.2) | 0.6 (1.3)
  Post-Intervention | 1.3 (1.1) | 0.9 (2.2)
Statistical Analysis 1: Comparison: Integrative Body Mind Training (IBMT) vs Relaxation Training (RT); Test type: Superiority; p = 0.03, threshold-free cluster enhancement — Threshold p<0.05

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Integrative Body Mind Training (IBMT) | Relaxation Training (RT)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-03-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT04261504/Prot_SAP_ICF_000.pdf